CLINICAL TRIAL: NCT06475365
Title: The Effect of Salt Water Gargling on Swallowing Dysfunction Following Multi-Level Anterior Cervical Discectomy and Fusion (ACDF): A Randomized Control Trial
Brief Title: Salt Water Gargling on Swallowing Following ACDF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Ram Alluri, Assistant Professor of Clinical Orthopaedic Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HS-24-00348
Record Dates: First submitted 2024-06-13; First posted 2024-06-26 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-03

CONDITIONS: Degeneration Spine; Cervical Radiculopathy; Cervical Stenosis; Cervical Spondylosis; Cervical Myelopathy; Dysphagia
Keywords: ACDF; Anterior cervical discectomy & fusion; Cervical spine; Dysphagia
MeSH Terms: conditions — Radiculopathy; Spondylosis; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Control (no intervention) & experimental (intervention). Both study arms will complete three (3) questionnaires at specified time points. In addition to questionnaires, the experimental group will receive an intervention of gargling warm salt water thrice daily (t.i.d.).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): This arm will receive no intervention. The patients in this arm will only be asked to complete the questionnaires related to the study. They will only receive the care as prescribed by their physician and care teams.
- Salt Water Gargle (Experimental): After their surgery, this arm will receive "treatment." Patients will be asked to gargle with a warm sodium chloride (salt water) solution. Patients will gargle with 15mL (15cc) of a premade solution of salt water one time (q.d.) on postoperative day 0 (POD 0), and three times a day (t.i.d.) for the next seven (7) days following their surgery (POD 1 - POD 7). Patients will also be asked to complete a series of study-related questionnaires at specified time points.
  Interventions: Other: Sodium chloride gargle

INTERVENTIONS:
Other: Sodium chloride gargle — 15mL salt water gargle
  Other Names: Salt water gargle
  Arms: Salt Water Gargle

SUMMARY:
The goal of this randomized control trial is to collect sufficient preliminary data on the efficacy of sodium chloride, hereafter referred to as "saltwater" or "saline" in reducing the difficulty of swallowing following multi-level anterior cervical discectomy and fusion (ACDF) procedures. The study population will consist of generally healthy adults ages 18 - 80. The main question it aims to answer is:

If the symptomatology and severity of swallowing difficulties following ACDF surgery can be reduced by gargling with warm salt water.

Researchers will compare the control and interventional arms to see if the proposed intervention of gargling with warm salt water improves difficulty swallowing following surgery.

Patients in the control arm will be asked to:

- Complete three (3) questionnaires at specified intervals (preoperative, postoperative day (POD) 1, 2, and 7; and at 1-month postoperatively).

Patients in the experimental/interventional arm will be asked to:

* Complete three (3) questionnaires at specified intervals (preoperative, postoperative day (POD) 1, 2, and 7; and at 1-month postoperatively).
* Gargle with a warm saltwater solution once on POD 0, and thrice daily from POD 1 to POD 7.

DETAILED DESCRIPTION:
Background & Hypothesis:

Dysphagia, or difficulty swallowing, often signifies structural or functional abnormalities in any of the three phases of swallowing and contributes to higher self-reported disability and lower physical health status. Dysphagia is a common postoperative complication following anterior cervical discectomy and fusion (ACDF) procedures. While most experience mild and transient symptoms, some individuals endure severe dysphagia, leading to significant postoperative morbidity.

Several studies have demonstrated the efficacy of corticosteroids administered intraoperatively during ACDF procedures. One prospective, randomized, double-blinded study, showed favorable results with local corticosteroid administration, resulting in a significant decrease in dysphagia during the immediate postoperative period to 1-month postoperatively. Although other studies have also reported favorable outcomes with corticosteroid use, they are still associated with considerable risks of adverse events. Corticosteroids have been linked to a higher incidence of postoperative infection, impairment of wound healing, and a 2- to 5-fold increase in wound complications across a variety of surgical specialties.

Salt water, also known as saline is associated with anti-inflammatory, anti-bacterial, and wound healing properties. Warm salt water rinses offer a more accessible, cost-effective alternative to corticosteroids, without their associated adverse effects. The study aims to investigate the efficacy of gargling salt water in reducing the severity and symptoms of swallowing difficulties following multi-level ACDF procedures.

This study is a single-center, prospective, randomized control trial. Only patients ≥ 18 years of age who are undergoing a multi-level (2-, 3-, or 4-level ACDF) and meet the general inclusion criterion will be invited to participate in the study.

Methodology:

1. Patients will be screened using the general inclusion/exclusion parameters
2. Patients will be randomized into one of two groups: control or experimental using a 1:1 ratio
3. Patients will complete three (3) questionnaires at selected time points throughout the study duration
4. Patients in the experimental arm will be asked to gargle with a saltwater solution one (1) time on POD 0 and three (3) times per day with approximately 15 milliliters (mL) per mouthful for seven (7) days (POD 1 - POD 7) + scheduled questionnaires
5. Patients in the control arm will only be asked to complete the scheduled questionnaires

Required questionnaires:

1. Swallow Quality of Life Questionnaire (SWAL-QOL)
2. Visual Analogue Scale - Neck (VAS Neck)
3. Eating Assessment Tool (EAT-10)

General study execution:

Patients in the interventional arm will be provided with a premade sodium chloride (sterile saltwater solution), 8-ounce-marked measuring cups, and a detailed instruction sheet with the relevant contacts for the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Patients undergoing a multi-level (2-, 3-, or 4-level) ACDF procedure
* Single-approach (anterior only) ACDF - English or Spanish-speaking patients
* Undergoing treatment at Keck Medical Center of USC

Exclusion Criteria:

* Patients ≤ 18 years of age
* Patients undergoing any revision ACDF procedure
* Patients undergoing ACDF with combined approaches (i.e. anterior + posterior)
* Patients with spinal pathologies or deformities that are non-degenerative or idiopathic (i.e. trauma, infection, malignancy, or tumor)
* Patients with a prior diagnosis related to swallowing issues (i.e. esophagitis, Barrett's esophagus, Sjogren syndrome, multiple sclerosis (MS), or laryngitis)
* Patients with an American Society of Anesthesiologists (ASA) score ≥ 4

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a SWAL-QOL Score of Greater Than 14 | 0 - 1 month
  The Swallowing-Related Quality of Life (SWAL-QOL) questionnaire is a 44-question assessment that measures the severity of oropharyngeal dysphagia (difficulty swallowing) and the impact it has on quality of life. Patients with score of greater than or equal to 14 are indicative of have some sort of difficulty with swallowing. This will be used to assess if patients in the Salt Water Gargle arm (intervention) have any relief after completing the described intervention.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) Score of 30 to 100 | 0 - 1 month
  On the NDI, a scores of ranging from 30 - 100 are indicative of mild to severe disability with respect to function of the neck. This will be used to assess if there is a correlation between a high SWAL-QOL score and a high NDI score.

CONTACTS AND LOCATIONS:
Overall Officials: Ram K Alluri, M.D., Principal Investigator — Assistant Professor of Clinical Orthopaedic Surgery
Locations (1):
- Keck Medical Center of the University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adenikinju AS, Halani SH, Rindler RS, Gary MF, Michael KW, Ahmad FU. Effect of perioperative steroids on dysphagia after anterior cervical spine surgery: A systematic review. Int J Spine Surg. 2017 Mar 6;11(2):9. doi: 10.14444/4009. eCollection 2017. PMID 28377867
- [Background] Anderson KK, Arnold PM. Oropharyngeal Dysphagia after anterior cervical spine surgery: a review. Global Spine J. 2013 Dec;3(4):273-86. doi: 10.1055/s-0033-1354253. Epub 2013 Aug 30. PMID 24436882
- [Background] Campbell PG, Yadla S, Malone J, Zussman B, Maltenfort MG, Sharan AD, Harrop JS, Ratliff JK. Early complications related to approach in cervical spine surgery: single-center prospective study. World Neurosurg. 2010 Aug-Sep;74(2-3):363-8. doi: 10.1016/j.wneu.2010.05.034. PMID 21492571
- [Background] Collins JR, Veras K, Hernandez M, Hou W, Hong H, Romanos GE. Anti-inflammatory effect of salt water and chlorhexidine 0.12% mouthrinse after periodontal surgery: a randomized prospective clinical study. Clin Oral Investig. 2021 Jul;25(7):4349-4357. doi: 10.1007/s00784-020-03748-w. Epub 2021 Jan 3. PMID 33389135
- [Background] Cloney MB, Garcia RM, Smith ZA, Dahdaleh NS. The Effect of Steroids on Complications, Readmission, and Reoperation After Posterior Lumbar Fusion. World Neurosurg. 2018 Feb;110:e526-e533. doi: 10.1016/j.wneu.2017.11.030. Epub 2017 Nov 16. PMID 29155116
- [Background] Gupta S, Jain A, Singla M. Is saltwater mouth rinse as effective as chlorhexidine following periodontal surgery? Evid Based Dent. 2021 Dec;22(4):130-131. doi: 10.1038/s41432-021-0227-6. Epub 2021 Dec 16. PMID 34916636
- [Background] Huynh NC, Everts V, Leethanakul C, Pavasant P, Ampornaramveth RS. Rinsing with Saline Promotes Human Gingival Fibroblast Wound Healing In Vitro. PLoS One. 2016 Jul 21;11(7):e0159843. doi: 10.1371/journal.pone.0159843. eCollection 2016. PMID 27441729
- [Background] Kalb S, Reis MT, Cowperthwaite MC, Fox DJ, Lefevre R, Theodore N, Papadopoulos SM, Sonntag VK. Dysphagia after anterior cervical spine surgery: incidence and risk factors. World Neurosurg. 2012 Jan;77(1):183-7. doi: 10.1016/j.wneu.2011.07.004. Epub 2011 Nov 15. PMID 22155226
- [Background] Kim HJ, Alluri R, Stein D, Lebl D, Huang R, Lafage R, Bennett T, Lafage V, Albert T. Effect of Topical Steroid on Swallowing Following ACDF: Results of a Prospective Double-Blind Randomized Control Trial. Spine (Phila Pa 1976). 2021 Apr 1;46(7):413-420. doi: 10.1097/BRS.0000000000003825. PMID 33273438
- [Background] Liu FY, Yang DL, Huang WZ, Huo LS, Ma L, Wang H, Yang SD, Ding WY. Risk factors for dysphagia after anterior cervical spine surgery: A meta-analysis. Medicine (Baltimore). 2017 Mar;96(10):e6267. doi: 10.1097/MD.0000000000006267. PMID 28272237
- [Background] National Institute on Deafness and Other Communication Disorders (National Institutes of Health). Dysphagia. NIH Publication No. 10-4307. Bethesda, MD: NIH; October 2010. Available at: http://www.nidcd.nih.gov/health/voice/Pages/dysph.aspx.
- [Background] Oh LJ, Ong S, Ghozy S, Dmytriw AA, Zuccato J, Mobbs R, Phan K, Dibas M, Faulkner H. Dysphagia rates in single- and multiple-level anterior cervical discectomy and fusion surgery: a meta-analysis. J Spine Surg. 2020 Sep;6(3):581-590. doi: 10.21037/jss-20-506. PMID 33102895
- [Background] Tasiou A, Giannis T, Brotis AG, Siasios I, Georgiadis I, Gatos H, Tsianaka E, Vagkopoulos K, Paterakis K, Fountas KN. Anterior cervical spine surgery-associated complications in a retrospective case-control study. J Spine Surg. 2017 Sep;3(3):444-459. doi: 10.21037/jss.2017.08.03. PMID 29057356
- [Background] Yee TJ, Swong K, Park P. Complications of anterior cervical spine surgery: a systematic review of the literature. J Spine Surg. 2020 Mar;6(1):302-322. doi: 10.21037/jss.2020.01.14. PMID 32309668
- See also: NIH Dysphagia — https://www.nidcd.nih.gov/health/dysphagia